CLINICAL TRIAL: NCT03889418
Title: Opioid Treatment and Recovery Through a Safe Pain Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ochsner Health System (Other)
Collaborators: Tulane University School of Public Health and Tropical Medicine (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Eboni Price-Haywood, Medical Director, Ochsner Health System
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01DA045029-01 (NIH)
Record Dates: First submitted 2019-03-20; First posted 2019-03-26 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Depression; Opioid Use; Chronic Pain; Anxiety
MeSH Terms: conditions — Depression; Chronic Pain; Anxiety Disorders | interventions — MCC protocol

STUDY DESIGN:
Intervention Model Description: This proposal is a 4-year type 2 effectiveness-implementation hybrid stepped wedge cluster randomized control (cRCT) trial to evaluate a multi-component intervention to: electronic medical recorded (EMR)clinical decision support (CDS) guided care; and stepped opioid collaborative care model (CCM) to improve opioid management of primary care patients with chronic non-cancer pain. The stepped wedge cRCT design will allow us to examine the clinical impact of the intervention as the two components are implemented in a stepwise fashion across the health system. The EMR CDS guided care component went live in all primary care clinics as the health system's standard of practice in October 2017. The stepped opioid CCM component will require 15 months to scale up in 3-month intervals across five geographic regions of the health system in the state of Louisiana. We will randomize the order in which stepped opioid CCM becomes available in each region
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic medical recorded clinical decision support (Active Comparator): Usual care only
  Interventions: Behavioral: Electronic medical recorded clinical decision support [EMR CDS]
- stepped opioid collaborative care model (Active Comparator): Usual care AND collaborative care with behavioral health integration
  Interventions: Behavioral: Electronic medical recorded clinical decision support [EMR CDS]; Behavioral: Stepped opioid collaborative care model [CCM]

INTERVENTIONS:
Behavioral: Electronic medical recorded clinical decision support [EMR CDS] — The opioid management tool has quick links to the Opioid Risk Tool (ORT), health maintenance reminders for risk mitigation tasks (pain management agreements; urine drug screening; prescribing naloxone); Pain Scale and depression/anxiety screen. The frequency with which providers are prompted to complete mitigation tasks is based on patients' level of risk for aberrant drug behavior defined by the ORT score. Additionally, the EMR CDS flags patients as high risk if one of the following criteria are met: (1) co-prescriptions for benzodiazepines; (2) active diagnosis of substance abuse in the last 12 months; or (3) MEDD >=90 mg. The ORT score, morphine equivalent daily dose (MEDD), and hyperlinks to the Louisiana pharmacy drug monitoring program data are visible in the prescription writer. If MEDD >=90 mg, the calculated MEDD is displayed in red font to alert the prescribing provider of high dosage. An Epic banner appears in charts to alert providers of existing pain management agreements.
Behavioral: Stepped opioid collaborative care model [CCM] — The licensed clinical social worker (LCSW) will provide counseling services as indicated (behavioral activation, psychotherapy, crisis planning, facilitating connection to substance abuse counseling and treatment); meet weekly with the consulting psychiatrist for complex case review and care plan adjustments; and supervise the community health worker (CHW) case management and depression/anxiety care management activities. The CHW will update assets and barriers to recovery and self-management and help patients navigate community resources. The clinical pharmacist will review and reconcile active medication lists, assess medication side effects, drug interactions and adverse events; monitor analgesia; recommend algorithm based anti-depression medication titration as indicated. The consulting psychiatrist will directly co-manage patients with severe mental illness, substance abuse and complex medication regimens.
  Arms: stepped opioid collaborative care model

SUMMARY:
Opioid prescription drug abuse has become a major public health concern in the United States with mortality rates from fatal overdoses reaching epidemic proportions. This opioid crisis coincides with national efforts to improve management of chronic non-cancer pain. The net result, however, has been ever-growing increases in medical expenditures related to prescription costs and increased healthcare service utilization among opioid abusers. Healthcare provider prescribing pattern, especially among non-pain management specialists such as primary care, is a major factor. Louisiana is a major contributor to the epidemic with the 7th highest opioid prescribing rates accompanied by a 12% increase in fatal overdoses.

Providers are overdue for implementing safe opioid management strategies in primary care to combat the opioid crisis. Recent practice guidelines provide recommendations on what to do for safe prescribing of opioids, but they do not provide guidance on how to translate them into practice. Health systems must find ways to accelerate guideline adoption in primary care in the face of an overdose crisis. Research that examines a combination workflow- and provider-focused strategies are needed. Given the high prevalence of psychiatric disorders among patients with chronic non-cancer pain, care team expansion with integration of collaborative mental/behavioral health services may be the solution. Collaborative care can extend opioid management beyond standardized monitoring of risk factors for opioid misuse or abuse and set clear protocols for next steps in management.

This study is aligned with the National Institute on Drug Abuse's interest in health systems research that examines approaches to screening, assessment, prevention, diagnosis and treatment for prescription drug abuse. It will examine the primary care practice redesign of managing chronic non-cancer pain within a large health system whose 40+ Accountable Care Network-affiliated, adult primary care clinics may serve as an example for transforming opioid management in primary care practices across the country. This four-year type 2 effectiveness-implementation hybrid stepped wedge cluster randomized control trial is designed to compare the clinical and cost effectiveness of electronic medical record-based clinical decision support guided care versus additional integrated, stepped collaborative care for opioid management of primary care patients with chronic non-cancer pain (clinical pharmacist for medication management; licensed clinical social worker for cognitive behavioral therapy and community health worker care coordination); and to examine facilitators and barriers to implementing this multi-component intervention. Investigators anticipate that our study results will elucidate the role of technology versus care team optimization in changing provider opioid prescribing behaviors. Investigators further anticipate that results of our study will demonstrate that integrated mental/behavioral health care for opioid management of chronic non-cancer pain increases value-based care and leads to greater efficiencies in the way that care is delivered.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Have a primary care provider at any of the study clinics
3. Receiving chronic opioid prescriptions (3 of the prior 4 months) for chronic non-cancer pain
4. Have a diagnosis of depression or anxiety

Exclusion Criteria:

1. Age less than 18 years
2. Active cancer or undergoing cancer treatment
3. Chronic cancer-related pain
4. Having a terminal illness
5. Receiving hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Health System - Research Dept, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Price-Haywood EG, Robinson W, Harden-Barrios J, Burton J, Burstain T. Intelligent Clinical Decision Support to Improve Safe Opioid Management of Chronic Noncancer Pain in Primary Care. Ochsner J. 2018 Spring;18(1):30-35. PMID 29559866
- [Background] Price-Haywood EG, Burton J, Burstain T, Harden-Barrios J, Lefante J, Shi L, Jamison RN, Bazzano A, Bazzano L. Clinical Effectiveness of Decision Support for Prescribing Opioids for Chronic Noncancer Pain: A Prospective Cohort Study. Value Health. 2020 Feb;23(2):157-163. doi: 10.1016/j.jval.2019.09.2748. Epub 2019 Nov 22. PMID 32113620
- [Background] Price-Haywood EG, Burton J, Harden-Barrios J, Bazzano A, Lefante J, Shi L, Jamison RN. Depression, anxiety, pain and chronic opioid management in primary care: Type II effectiveness-implementation hybrid stepped wedge cluster randomized trial. Contemp Clin Trials. 2021 Feb;101:106250. doi: 10.1016/j.cct.2020.106250. Epub 2020 Dec 14. PMID 33326877
- [Result] Price-Haywood EG, Burton JH, Harden-Barrios J, Bazzano A, Shi L, Lefante J, Jamison RN. Decision Support and Behavioral Health for Reducing High-Dose Opioids in Comorbid Chronic Pain, Depression and Anxiety: Stepped-Wedge Cluster Randomized Trial. J Gen Intern Med. 2024 Nov;39(15):2952-2960. doi: 10.1007/s11606-024-08965-7. Epub 2024 Aug 2. PMID 39095571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient ENROLLMENT was CONTINUOUS following the go-live dates for each health system geographic region. Participants were referred for collaborative care management (CCM) between April 2019 and December 2021 for eligibility screening. All enrollment was completed by January 2022. A propensity matched control group (usual care) was identified among patients receiving care within the health system during the time of this study who were never exposed to the collaborative care intervention.
Pre-assignment Details: Clinics within the same geographic region have the same operations management team and share resources. Using computer generated random numbers, each region (cluster) was randomized to the order of collaborative care intervention roll out in 5 steps occurring in 3 to 4-month intervals. Randomized sequence: (1) April 2019, Region 1; (2) July 2019, Region 2; (3) October 2019, Region 3; (4) January 2020, Region 4; (5) April 2020, Region 5.
Units Other Than Participants: Geographic region
Groups:
- Sequence 1: Electronic Medical Recorded Clinical Decision Support (EMR-CDS): Usual care group within Region 1 of the health system that was only exposed to EMR-CDS for chronic opioid management.
- Sequence 1: Stepped Opioid Collaborative Care Management (EMR-CDS With CCM): Study group in Region 1 of the health system who received usual care (EMR-CDS) AND collaborative care management with behavioral health integration.
- Sequence 2: EMR-CDS: Study group in Region 2 of health system receiving usual care
- Sequence 2: EMR-CDS With CCM: Study group in Region 2 of the health system receiving EMR-CDS and CCM
- Sequence 3: EMR-CDS: Study group in Region 3 of health system receiving usual care
- Sequence 3: EMR-CDS With CCM: Study group in Region 3 of the health system receiving EMR-CDS and CCM
- Sequence 4: EMR-CDS: Study group in Region 4 of health system receiving usual care
- Sequence 4: EMR With CCM: Study group in Region 4 of the health system receiving EMR-CDS and CCM
- Sequence 5: EMR-CDS: Study group in Region 5 of health system receiving usual care
- Sequence 5: EMR With CCM: Study group in Region 5 of the health system receiving EMR-CDS and CCM
Period: April-June 2019 (Months 0-3)
Arm/Group | Sequence 1: Electronic Medical Recorded Clinical Decision Support (EMR-CDS) | Sequence 1: Stepped Opioid Collaborative Care Management (EMR-CDS With CCM) | Sequence 2: EMR-CDS | Sequence 2: EMR-CDS With CCM | Sequence 3: EMR-CDS | Sequence 3: EMR-CDS With CCM | Sequence 4: EMR-CDS | Sequence 4: EMR With CCM | Sequence 5: EMR-CDS | Sequence 5: EMR With CCM
Started ([EMR-CDS with CCM] participants started enrollment in region 1 in period 1. In Region 2, 3, 4 & 5, only EMR-CDS (usual care) matched controls were identified. Note: Number of participants to start a period includes number that completed the previous period and newly enrolled participants.) | 48; 1 Geographic region | 10; 1 Geographic region | 21; 1 Geographic region | 0; 0 Geographic region | 14; 1 Geographic region | 0; 0 Geographic region | 10; 1 Geographic region | 0; 0 Geographic region | 12; 1 Geographic region | 0; 0 Geographic region
Completed | 47; 1 Geographic region | 10; 1 Geographic region | 21; 1 Geographic region | 0; 0 Geographic region | 14; 1 Geographic region | 0; 0 Geographic region | 10; 1 Geographic region | 0; 0 Geographic region | 12; 1 Geographic region | 0; 0 Geographic region
Not Completed | 1; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: July-September 2019 (Months 4-6)
Arm/Group | Sequence 1: Electronic Medical Recorded Clinical Decision Support (EMR-CDS) | Sequence 1: Stepped Opioid Collaborative Care Management (EMR-CDS With CCM) | Sequence 2: EMR-CDS | Sequence 2: EMR-CDS With CCM | Sequence 3: EMR-CDS | Sequence 3: EMR-CDS With CCM | Sequence 4: EMR-CDS | Sequence 4: EMR With CCM | Sequence 5: EMR-CDS | Sequence 5: EMR With CCM
Started ([EMR-CDS with CCM] participants started enrollment in region 2 in period 2. In Region 3, 4 & 5, only EMR-CDS (usual care) matched controls were identified. Note: Number of participants to start a period includes number that completed the previous period and newly enrolled participants.) | 54; 1 Geographic region | 20; 1 Geographic region | 23; 1 Geographic region | 2; 1 Geographic region | 16; 1 Geographic region | 1; 0 Geographic region | 10; 1 Geographic region | 0; 0 Geographic region | 13; 1 Geographic region | 0; 0 Geographic region
Completed | 54; 1 Geographic region | 19; 1 Geographic region | 22; 1 Geographic region | 2; 1 Geographic region | 16; 1 Geographic region | 1; 0 Geographic region | 10; 1 Geographic region | 0; 0 Geographic region | 13; 1 Geographic region | 0; 0 Geographic region
Not Completed | 0; 0 Geographic region | 1; 0 Geographic region | 1; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: October-December 2019 (Month 7-9)
Arm/Group | Sequence 1: Electronic Medical Recorded Clinical Decision Support (EMR-CDS) | Sequence 1: Stepped Opioid Collaborative Care Management (EMR-CDS With CCM) | Sequence 2: EMR-CDS | Sequence 2: EMR-CDS With CCM | Sequence 3: EMR-CDS | Sequence 3: EMR-CDS With CCM | Sequence 4: EMR-CDS | Sequence 4: EMR With CCM | Sequence 5: EMR-CDS | Sequence 5: EMR With CCM
Started ([EMR-CDS with CCM] participants started enrollment in region 3 in period 3. In Regions 4 & 5, EMR-CDS (usual care) matched controls were identified. Note: Number of participants to start a period includes number that completed the previous period and newly enrolled participants.) | 60; 1 Geographic region | 36; 1 Geographic region | 28; 1 Geographic region | 11; 1 Geographic region | 16; 1 Geographic region | 1; 1 Geographic region | 12; 1 Geographic region | 0; 0 Geographic region | 16; 1 Geographic region | 1; 0 Geographic region (Patient recruited out of sequence but retained in study.)
Completed | 60; 1 Geographic region | 36; 1 Geographic region | 28; 1 Geographic region | 11; 1 Geographic region | 16; 1 Geographic region | 1; 1 Geographic region | 12; 1 Geographic region | 0; 0 Geographic region | 15; 1 Geographic region | 1; 0 Geographic region
Not Completed | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 1; 0 Geographic region | 0; 0 Geographic region
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: January - March 2020 (Month 10-12)
Arm/Group | Sequence 1: Electronic Medical Recorded Clinical Decision Support (EMR-CDS) | Sequence 1: Stepped Opioid Collaborative Care Management (EMR-CDS With CCM) | Sequence 2: EMR-CDS | Sequence 2: EMR-CDS With CCM | Sequence 3: EMR-CDS | Sequence 3: EMR-CDS With CCM | Sequence 4: EMR-CDS | Sequence 4: EMR With CCM | Sequence 5: EMR-CDS | Sequence 5: EMR With CCM
Started ([EMR-CDS with CCM] participants started enrollment in region 4 in period 4. In Region 5, only EMR-CDS (usual care) matched controls were identified. Note: Number of participants to start a period includes number that completed the previous period and newly enrolled participants.) | 67; 1 Geographic region | 48; 1 Geographic region | 34; 1 Geographic region | 24; 1 Geographic region | 16; 1 Geographic region | 2; 1 Geographic region | 13; 1 Geographic region | 5; 1 Geographic region | 16; 1 Geographic region | 1; 0 Geographic region
Completed | 67; 1 Geographic region | 48; 1 Geographic region | 34; 1 Geographic region | 23; 1 Geographic region | 16; 1 Geographic region | 2; 1 Geographic region | 13; 1 Geographic region | 3; 1 Geographic region | 16; 1 Geographic region | 1; 0 Geographic region
Not Completed | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 1; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 2; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Period: April - June 2020 (Month 13-15)
Arm/Group | Sequence 1: Electronic Medical Recorded Clinical Decision Support (EMR-CDS) | Sequence 1: Stepped Opioid Collaborative Care Management (EMR-CDS With CCM) | Sequence 2: EMR-CDS | Sequence 2: EMR-CDS With CCM | Sequence 3: EMR-CDS | Sequence 3: EMR-CDS With CCM | Sequence 4: EMR-CDS | Sequence 4: EMR With CCM | Sequence 5: EMR-CDS | Sequence 5: EMR With CCM
Started ([EMR-CDS with CCM] participants started enrollment in region 5 in period 5. Note: Number of participants to start a period includes number that completed the previous period and newly enrolled participants.) | 75; 1 Geographic region | 60; 1 Geographic region | 38; 1 Geographic region | 27; 1 Geographic region | 19; 1 Geographic region | 2; 1 Geographic region | 16; 1 Geographic region | 3; 1 Geographic region | 19; 1 Geographic region | 4; 1 Geographic region
Completed | 75; 1 Geographic region | 59; 1 Geographic region | 38; 1 Geographic region | 26; 1 Geographic region | 19; 1 Geographic region | 2; 1 Geographic region | 16; 1 Geographic region | 3; 1 Geographic region | 19; 1 Geographic region | 4; 1 Geographic region
Not Completed | 0; 0 Geographic region | 1; 0 Geographic region | 0; 0 Geographic region | 1; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: July 2020 - January 2022 (Month 16-28)
Arm/Group | Sequence 1: Electronic Medical Recorded Clinical Decision Support (EMR-CDS) | Sequence 1: Stepped Opioid Collaborative Care Management (EMR-CDS With CCM) | Sequence 2: EMR-CDS | Sequence 2: EMR-CDS With CCM | Sequence 3: EMR-CDS | Sequence 3: EMR-CDS With CCM | Sequence 4: EMR-CDS | Sequence 4: EMR With CCM | Sequence 5: EMR-CDS | Sequence 5: EMR With CCM
Started | 101; 1 Geographic region | 112; 1 Geographic region | 67; 1 Geographic region | 52; 1 Geographic region | 21; 1 Geographic region | 6; 1 Geographic region | 24; 1 Geographic region | 21; 1 Geographic region | 23; 1 Geographic region | 42; 1 Geographic region
Completed | 100; 1 Geographic region | 108; 1 Geographic region | 63; 1 Geographic region | 50; 1 Geographic region | 21; 1 Geographic region | 6; 1 Geographic region | 24; 1 Geographic region | 19; 1 Geographic region | 23; 1 Geographic region | 38; 1 Geographic region
Not Completed | 1; 0 Geographic region | 4; 0 Geographic region | 4; 0 Geographic region | 2; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 0; 0 Geographic region | 2; 0 Geographic region | 0; 0 Geographic region | 4; 0 Geographic region
Not completed — Death | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 4 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Electronic Medical Recorded Clinical Decision Support: Electronic medical recorded clinical decision support (usual care)
- Total: Total of all reporting groups
Arm/Group | Electronic Medical Recorded Clinical Decision Support | Stepped Opioid Collaborative Care Model | Total
Number analyzed (Participants) | 239 | 239 | 478
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (14.8) | 57.3 (11.9) | 56.6 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 169 | 341
  Male | 67 | 70 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 226 | 231 | 457
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 85 | 89 | 174
  White | 152 | 148 | 300
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 239 | 239 | 478
Insurance Type [Count of Participants; unit: Participants]
  Commercial | 107 | 127 | 234
  Medicare | 104 | 93 | 197
  Medicaid | 20 | 16 | 36
  Self-Pay or Uninsured | 5 | 3 | 8
  Unknown | 3 | 0 | 3
Charlson Comorbidity Index [Mean (Standard Deviation); unit: Score on a scale] — Charlson Comorbidity Index is a validated method of estimating the 10-year risk of death from concurrent disease. The higher the score, the higher the predicted risk of mortality. The index score is based on 17 different medical conditions categories defined by the International Classification of Disease. Each comorbidity category has an associated weight (from 1 to 6). The condition-specific scores are summed for the overall score (range 0 to 29). Refer to online calculators to predict mortality risk for a given score.
  Score on a scale | 4.0 (3.1) | 4.1 (3.4) | 4.1 (3.3)
Depression [Count of Participants; unit: Participants] — International Classification Disease diagnose code for Major Depression Disorder documented in patient medical record
  Participants | 221 | 224 | 445
Anxiety [Count of Participants; unit: Participants] — International Classification Disease diagnosis code for anxiety disorders documented in patient medical record
  Participants | 208 | 206 | 414
Morphine Equivalent Daily Dose [Mean (Standard Deviation); unit: mg per day] — Morphine Equivalent Daily Dose (MEDD) is calculated by determining the total daily amount of a prescribed opioid, multiplying the dose of the opioid by a conversion factor to ascertain morphine milligram equivalents and then adding up the dosage. Population: Only patients who survived throughout the study time period and with data documented in the electronic medical record system 12-months before the index date are included in the analysis.
  mg per day
    number analyzed (Participants) | 231 | 221 | 452
    (all) | 40.3 (48.9) | 50.9 (73.2) | 45.5 (62.5)

OUTCOME MEASURES:

1. Primary Outcome: Odds of Morphine Equivalent Daily Dose (MEDD) of Opioid Prescription >=50 mg
Description: Participants' opioid medication orders were monitored for 12 months prior to and following entry into study (index event). This outcome represents the odds of having an average MEDD ≥ 50 mg in the pre-index and post-index periods for the collaborative care and usual care groups. Odds of an event is defined as the ratio of the probability that the event will happen (prescribed high dose opioid) to the probability that the event will not happen (not prescribed high dose opioid)
Time Frame: 12 months prior to index event (pre-index period) and 12 months following index event (post-index period)
Population: All participants who survived through end of study and had at least one documented opioid medication order, excluding buprenorphine and methadone, in the 12-month pre-index period are included in the analysis. Patients who died during the course of the study or were missing prescription data at baseline are not included in this analysis.
Measure: Number (95% Confidence Interval); unit: odds of prescription high dose
Arm/Group | Electronic Medical Recorded Clinical Decision Support | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 231 | 221
odds of prescription high dose
  Pre-Index | 0.209 [0.149 to 0.295] | 0.417 [0.312 to 0.557]
  Post-Index | 0.185 [0.129 to 0.264] | 0.364 [0.270 to 0.491]
Statistical Analysis 1: Comparison: Electronic Medical Recorded Clinical Decision Support vs Stepped Opioid Collaborative Care Model; Test type: Superiority; p = 0.956, Mixed Models Analysis; Odds Ratio, log = -0.009, 95% CI 2-sided [-0.309 to 0.292], Standard Error of Mean 0.153

2. Secondary Outcome: Rate Ratios for Average Morphine Equivalent Daily Dose (MEDD) of Opioid Prescriptions in the Post-index Versus Pre-index Periods
Description: Participants' opioid medication orders were monitored for 12 months prior to and following entry into study (index event). This outcome represents the rate ratio of average MEDD in the post-index versus pre-index periods for the Behavioral Collaborative Care (BHI-CCM + EMR-CDS) and Usual Care (EMR-CDS only) groups. The rate ratio compares the average dose of opioid prescription in the post-index period to the pre-index period. A rate ratio less than 1 indicates that the average dose decreased.
Time Frame: 12 months prior to index event (pre-index period) and 12 months following index event (post-index period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Rate Ratio of average opioid dose
Arm/Group | Electronic Medical Recorded Clinical Decision Support | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 231 | 221
Rate Ratio of average opioid dose | 0.957 [0.903 to 1.014] | 0.863 [0.798 to 0.934]
Statistical Analysis 1: Comparison: Electronic Medical Recorded Clinical Decision Support vs Stepped Opioid Collaborative Care Model; Test type: Superiority; p = 0.039, Mixed Models Analysis; Risk Ratio, log = -0.103, 95% CI 2-sided [-0.200 to -.005], Standard Error of Mean 0.050

3. Secondary Outcome: Inpatient Hospital Admission Per 1000 Participants
Description: Participants' non-elective inpatient hospital admissions were monitored for 12 months prior to and following date of enrollment in study. This outcome represents the number of admissions in the pre-index and post-index periods for the study groups
Time Frame: 12 months prior to index event (pre-index period) and 12 months following index event (post-index period)
Population: All participants who died during the course of the study are excluded from the analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: Admissions per 1000 participants
Arm/Group | Electronic Medical Recorded Clinical Decision Support | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 235 | 236
Admissions per 1000 participants
  Pre-Index | 528 [362 to 769] | 309 [213 to 450]
  Post-Index | 413 [276 to 616] | 254 [170 to 379]
Statistical Analysis 1: Comparison: Electronic Medical Recorded Clinical Decision Support vs Stepped Opioid Collaborative Care Model; Test type: Superiority; p = 0.864, Mixed Models Analysis; Rate Ratio, log = 0.049, 95% CI 2-sided [-0.506 to 0.603], Standard Error of Mean 0.282

4. Secondary Outcome: Emergency Department Visits Per 1000 Participants
Description: Participants' emergency department (ED) visits were monitored for 12 months prior to and following date of enrollment in study. This outcome represents the number of ED visits in the pre-index and post-index periods for the study groups
Time Frame: 12 months prior to index event (pre-index period) and 12 months following index event (post-index period)
Population: All participants who died during the course of the study are excluded from the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Visits per 1000 participants
Arm/Group | Electronic Medical Recorded Clinical Decision Support | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 235 | 236
Visits per 1000 participants
  Pre-Index | 1626 [1243 to 2127] | 1352 [1034 to 1767]
  Post-Index | 1526 [1131 to 2059] | 1292 [958 to 1742]
Statistical Analysis 1: Comparison: Electronic Medical Recorded Clinical Decision Support vs Stepped Opioid Collaborative Care Model; Test type: Superiority; p = 0.901, Mixed Models Analysis; rate ratio, log = 0.018, 95% CI 2-sided [-0.272 to 0.308], Standard Error of Mean 0.148

5. Secondary Outcome: Proportion of Patients Exposed to Collaborative Care With Improvement in Symptoms of Depression
Description: Participants in the collaborative care group were administered the Patient Health Questionnaire (PHQ)-9 questionnaire at baseline and every 4 weeks following date of enrollment in study. The PHQ-9 is a nine item questionnaire. The total score ranges from 0 to 27 (scores of 5-9 mild depression; 10-14 moderate depression; 15-19 moderately severe depression; ≥ 20 severe depression). This single-group outcome represents the number of participants who entered the study with symptoms of moderate to severe depression (PHQ-9 score ≥ 10) and achieved a PHQ-9 score < 10 on the last completed questionnaire.
Time Frame: 12 months following index event (post-index period)
Population: All participants in the collaborative care arm of the study with a baseline PHQ-9 score ≥ 10 who completed at least two questionnaires and survived through end of study were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 209
Participants | 129

6. Secondary Outcome: Proportion of Patients Exposed to Collaborative Care With Improvement in Symptoms of Anxiety
Description: Participants in the collaborative care group were administered the Generalized Anxiety Disorder (GAD)-7 questionnaire at baseline and every 4 weeks following date of enrollment in study. The GAD-7 is a seven item questionnaire. The total score ranges from 0 to 21 (scores of 5-9 mild anxiety; 10-14 moderate anxiety; 15-21 severe anxiety).This single-group outcome represents the number of participants who entered the study with symptoms of moderate to severe anxiety (GAD-7 score ≥ 10) and achieved a GAD-7 score < 10 on the last completed questionnaire
Time Frame: 12 months following index event (post-index period)
Population: All participants in the collaborative care study group with a baseline GAD-7 score ≥ 10 who completed at least two questionnaires and survived through end of study were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 161
Participants | 92

7. Secondary Outcome: Change in Patient Rating of Quality of Life
Description: Participants in the Collaborative Care group were administered the Patient Reported Outcomes Measurement Information System (PROMIS) 10 item questionnaire at baseline and every 12 weeks following enrollment in study. A PROMIS score of 50 is the average (or mean) score for the U.S. general population. This single-group outcome represents the average change in PROMIS-10 global mental health score from the first to the last completed questionnaire during the acute phase.
Time Frame: Baseline, 12-months following index event (post-index period)
Population: All Collaborative Care participants who completed at least two questionnaires and survived through end of study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 217
units on a scale
  Baseline PROMIS-10 Global Mental Health Score | 34.001 (7.191)
  Change in PROMIS-10 Global Mental Health Score | 2.000 (6.730)
  Baseline PROMIS-10 Global Physical Health Score | 35.815 (5.625)
  Change in PROMIS-10 Global Physical Health Score | 0.929 (5.275)

8. Secondary Outcome: Change in the Average Pain Score Among Participants Exposed to Collaborative Care
Description: Participants in the collaborative care group were administered the Pain Enjoyment of Life General Activity (PEG)-3 questionnaire at baseline and every 4 weeks during the acute phase of treatment. THE PEG-3 consists of 3 questions - each with a rating scale 0 (no pain; no interference) to 10 (worse pain; completely interferes). The score is generated by summing the score of the 3 scales (max 30 points) and then dividing by 3. The measure is reliable with construct validity and responsive among primary care patients. This single-group outcome represents the average change in PEG-3 score from the first to the last completed questionnaire during the acute phase.
Time Frame: 12 months following index event (post-index period)
Population: All participants in the collaborative care study group who completed at least two questionnaires and survived through end of study were included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 199
score on a scale
  Baseline score | 6.5 (1.7)
  Average change in score | -1.3 (1.8)

9. Secondary Outcome: New Post-index Documentation for Signed Pain Management Agreement (Pain Contract)
Description: Participants' pain contracts were monitored for 12 months prior to and following date of enrollment in study. This outcome represents the number of participants with a documented pain contract in the post-index period among those with no pain contract in the pre-index period
Time Frame: 12 months following index event (post-index period)
Population: Participants who survived through end of study and had no documented pain contract in the 12 months prior to enrollment in study were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Electronic Medical Recorded Clinical Decision Support | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 183 | 188
Participants | 21 | 23

10. Secondary Outcome: New Post-index Order for Urine Drug Screen (UDS)
Description: Participants' UDS were monitored for 12 months prior to and following date of enrollment in study. This outcome represents the number of participants with a documented UDS order in the post-index period among those with no UDS order in the pre-index period
Time Frame: 12 months following index event (post-index period)
Population: All participants who survived through end of study or loss to follow-up and had no documented UDS order in the 12 months prior to enrollment in study
Measure: Count of Participants; unit: Participants
Arm/Group | Electronic Medical Recorded Clinical Decision Support | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 160 | 149
Participants | 23 | 33

11. Secondary Outcome: New Post-index Naloxone Prescription Order
Description: Participants' medication orders were monitored for 12 months prior to and following date of enrollment in study. This outcome represents the number of participants with naloxone orders in the post-index period among those with no naloxone orders in the pre-index period
Time Frame: 12 months following index event (post-index period)
Population: Participants who did not naloxone orders documented in their medical record in the 12 months prior to enrollment in study OR who survived to the end of the study were included from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Electronic Medical Recorded Clinical Decision Support | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 222 | 199
Participants | 10 | 23

12. Secondary Outcome: Change in Rate of Patient Report of Opioid Misuse
Description: Change in Current Opioid Misuse Measure-9 (COMM-9) scores: The COMM-9 is a 9-item questionnaire with a 5-item response scale (0=never; 4=very often) that captures a 30-day period and only includes behaviors that can change over time (score range 0 to 36). Scoring greater than 4 are identified as being at risk for medication misuse. Participants in the Collaborative Care group were administered the COMM-9 questionnaire at baseline and every 4 weeks during the acute phase of treatment. This single-group outcome represents the average change in COMM-9 score from the first to the last completed questionnaire during the acute phase.
Time Frame: Baseline, 12 months following index event (post-index period)
Population: All collaborative care participants who completed at least two questionnaires and survived through end of study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 145
units on a scale
  Baseline score | 4.8 (2.9)
  Average change in score | -1.1 (2.6)

13. Secondary Outcome: New Post-index Documentation for Referral to Any Non-mental/Behavioral Health Specialty Service
Description: Participants' non-mental/behavioral health specialty service referrals (e.g. physical therapy, orthopedics) were monitored for 12 months prior to and following date of enrollment in study. This outcome represents the number of participants with referrals in the post-index period among those with no referrals in the pre-index period
Time Frame: 12 months following index event (post-index period)
Population: All participants who survived through end of study and had no documented referrals to non-mental/behavioral health specialty services in the 12 months prior to enrollment in study were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Electronic Medical Recorded Clinical Decision Support | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 115 | 85
Participants | 40 | 45

14. Secondary Outcome: New Post-index Orders for Antidepressant Medications
Description: Participants' medication orders were monitored for 12 months prior to and following date of enrollment in study. This outcome represents the number of participants with a new order for antidepressants in the post-index period among those with no orders in the pre-index period
Time Frame: 12 months following index event (post-index period)
Population: All participants who survived through end of study and had no orders for antidepressants in the 12 months prior to enrollment in study were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Electronic Medical Recorded Clinical Decision Support | Stepped Opioid Collaborative Care Model
Number analyzed (Participants) | 117 | 98
Participants | 37 | 49

15. Secondary Outcome: Provider Experience With Managing Depression/Anxiety/Pain
Description: Provider ratings of their experience with managing depression/anxiety/pain
Time Frame: Baseline
Population: A cross-sectional survey was administered to primary care providers in December 2019 for baseline measure of provider confidence in managing depression, anxiety and chronic pain and use of defined care management protocols when prescribing medications. 93 out of 226 (41%) providers responded to the survey.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Care Providers: Physicians and Advanced Practice Practitioners who provide primary care within the health system
Arm/Group | Primary Care Providers
Number analyzed (Participants) | 93
Participants
  Confident in ability to manage depression or anxiety: Strongly Agree or Agree | 83
  Confident in ability to manage depression or anxiety: Neutral/Disagree/Strongly Disagree | 10
  Confident in ability to manage depression or anxiety: Missing Data | 0
  Use care management protocol when depression or anxiety medication prescribed: Strongly Agree or Agree | 45
  Use care management protocol when depression or anxiety medication prescribed: Neutral/Disagree/Strongly Disagree | 47
  Use care management protocol when depression or anxiety medication prescribed: Missing Data | 1
  Confident in ability to manage chronic pain: Strongly Agree or Agree | 21
  Confident in ability to manage chronic pain: Neutral/Disagree/Strongly Disagree | 70
  Confident in ability to manage chronic pain: Missing Data | 2
  Use care management protocol when opioid medications prescribed: Strongly Agree or Agree | 44
  Use care management protocol when opioid medications prescribed: Neutral/Disagree/Strongly Disagree | 48
  Use care management protocol when opioid medications prescribed: Missing Data | 1

ADVERSE EVENTS:
Time Frame: Using Diagnosis Related Group (DRG) codes, adverse events were assessed during 12 months following index event
Description: Serious Adverse Events include inpatient admissions with emergency or non-elective admission types with a length of stay >1 day.
Arm/Group | Electronic Medical Recorded Clinical Decision Support | Stepped Opioid Collaborative Care Model
All-Cause Mortality (participants affected / at risk) | 4/239 | 3/239
Serious Adverse Events (participants affected / at risk) | 39/239 | 35/239
Other Adverse Events (participants affected / at risk) | 24/239 | 17/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electronic Medical Recorded Clinical Decision Support (N=239) | Stepped Opioid Collaborative Care Model (N=239)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Amputation (Surgical and medical procedures) | 2 (2) | 1 (1)
Atherosclerosis (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Complications of treatment (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes (Endocrine disorders) | 4 (4) | 0 (0)
Disorders of pancreas except malignancy (Gastrointestinal disorders) | 1 (1) | 1 (1)
Epistaxis (General disorders) | 1 (1) | 0 (0)
Esophagitis, Gastroenteritis and Misc Digestive Disorders (Gastrointestinal disorders) | 1 (1) | 2 (2)
Operating Room Procedure (Surgical and medical procedures) | 3 (4) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 5 (10) | 5 (5)
Hip and femur procedure (Surgical and medical procedures) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 1 (6) | 0 (0)
Infectious and parasitic diseases (Infections and infestations) | 2 (2) | 0 (0)
Intracranial hemorrhage or cerebral infarction (Nervous system disorders) | 1 (1) | 2 (2)
Kidney and urinary tract infections (Renal and urinary disorders) | 0 (0) | 1 (1)
Major chest trauma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Major gastrointestinal disorders and peritoneal infections (Gastrointestinal disorders) | 1 (1) | 0 (0)
Major hematological and immunological diagnoses (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Major small and large bowel procedures (Gastrointestinal disorders) | 0 (0) | 1 (1)
Medical back problems (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Minor skin disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Disorders of nutrition, metabolism, fluids and electrolytes (Endocrine disorders) | 3 (4) | 1 (1)
Other kidney and urinary tract diagnoses (Renal and urinary disorders) | 2 (3) | 0 (0)
Other skin, subcutaneous tissue and breast procedures (Surgical and medical procedures) | 2 (2) | 1 (1)
Other vascular procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Peritoneal adhesiolysis (Surgical and medical procedures) | 1 (1) | 0 (0)
Post-operative and post-traumatic infections (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary edema and respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Red blood cell disorder (Blood and lymphatic system disorders) | 4 (20) | 3 (10)
Renal failure (Renal and urinary disorders) | 4 (4) | 1 (1)
Respiratory infections and inflammations (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Respiratory system diagnosis with ventilator support (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Seizures (Nervous system disorders) | 1 (1) | 1 (1)
Septicemia or severe sepsis (Infections and infestations) | 1 (1) | 8 (9)
Simple pneumonia and pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Skin graft (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Spinal procedures or spinal neurostimulators (Surgical and medical procedures) | 0 (0) | 1 (1)
Syncope and collapse (Nervous system disorders) | 1 (1) | 0 (0)
Tracheostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Traumatic stupor and coma (Nervous system disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electronic Medical Recorded Clinical Decision Support (N=239) | Stepped Opioid Collaborative Care Model (N=239)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 24 (33) | 17 (32)

LIMITATIONS AND CAVEATS:
All data collected for the study were extracted from the health system electronic medical system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT03889418/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT03889418/SAP_001.pdf